CLINICAL TRIAL: NCT02656238
Title: New International CTEPH Database
Status: Completed | Type: Observational
Sponsor: International CTEPH Association (Other)
Responsible Party: Sponsor
Other Study IDs: CTEPH Registry
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; CTEPH
Keywords: CTEPH; Balloon pulmonary angioplasty; Chronic thromboembolic pulmonary hypertension; Pulmonary endarterectomy; BPA; PEA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The New International CTEPH Database is a prospective, observational multi-center disease registry run by the International CTEPH Association (ICA), which will collect data in chronic thromboembolic pulmonary hypertension (CTEPH) patients worldwide. The registry will run for approximately 5 years. Its objective is to provide an overview on epidemiology of CTEPH, mode of diagnosis and treatment approaches worldwide as well as determinants of long-term outcomes as measured by New York Heart Association (NYHA) functional class and survival.

The data collected will improve the knowledge and understanding of this condition, support the further development of diagnosis and treatment guidelines for patients with CTEPH, and contribute to improving patient care in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with chronic thromboembolic pulmonary hypertension (CTEPH) (incident patients)
* Patients must have been treated with anti-coagulation for at least 3 months before diagnosis of CTEPH
* Patients must be willing to provide informed consent
* Patients must meet the following criteria for CTEPH:

  * Mean pulmonary artery pressure (PAP) ≥ 25 mmHg at rest
  * Abnormal VQ scan, pulmonary angiogram, computed tomography (CT) pulmonary angiogram, or magnetic resonance (MR) pulmonary angiogram confirming chronic thromboembolic disease as recommended by standard guidelines

Exclusion Criteria:

* None specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients recently diagnosed with chronic thromboembolic pulmonary hypertension (CTEPH), meeting the registry's inclusion criteria, are eligible for inclusion into the New International CTEPH Database.
  Only newly diagnosed, i.e. incident patients are eligible for inclusion. A patient is considered an incident patient if a diagnostic heart catheterization was performed within 1 year prior to the initial inclusion visit (for the first patient included) at the site participating in the New International CTEPH Database.
Sampling Method: Non-Probability Sample
Enrollment: 1019 (Actual)
Dates: Start 2015-02; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Death | Min. 3 years
Lung transplantation | Min. 3 years
Change in New York Heart Association (NYHA) functional class | Min 3. years

SECONDARY OUTCOMES:
Age at diagnosis | Min. 3 years
Gender | Min. 3 years
Ethnicity | Min. 3 years
Disease severity | Min. 3 years
  As measured by New York Heart Association (NYHA) functional class
History of deep vein thrombosis (DVT) | Min. 3 years
History of acute pulmonary embolism | Min. 3 years
Hemodynamic parameters | Min. 3 years
Patient on oxygen (yes/no) | Min. 3 years
Medical treatment | Min. 3 years
  e.g. mono- versus combination therapy
Pulmonary endarterectomy (PEA) | Min. 3 years
  e.g. operated versus non-operated
Balloon pulmonary angioplasty (BPA) | Min. 3 years
  e.g. BPA versus pulmonary endarterectomy (PEA)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (3):
  - UC San Diego, La Jolla, California
  - University of Maryland, Baltimore, Maryland
  - Cleveland Clinic, Cleveland, Ohio
- Australia (2):
  - St Vincent's Hospital, Darlinghurst
  - The Alfred Hospital, Prahran
- University Clinics of Vienna, Vienna, Austria
- University Hospitals of Leuven, Leuven, Belgium
- Brazil (2):
  - Hospital São Paulo, Federal University of São Paulo, São Paulo
  - University of Sao Paulo Medical School, São Paulo
- Toronto General Hospital, Toronto, Ontario, Canada
- Aarhus University Hospital, Aarhus, Denmark
- Kasr Alaini School of Medicine, Cairo, Egypt
- Helsinki University Hospital, Helsinki, Finland
- Germany (3):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum des Saarlandes, Homburg
- University of Pavia, Pavia, Italy
- Japan (4):
  - Chiba University Hospital, Chiba
  - Kobe University Graduate School of Medicine, Kobe
  - National Hospital Organization Okayama, Okayama
  - Kyorin University Hospital, Tokyo
- VU University Medical Center, Amsterdam, Netherlands
- Poland (3):
  - Europejskim Centrum Zdrowia Otwock, Otwock
  - Medical University of Warsaw, Warsaw
  - Wojewódzki Szpital Specjalistyczny, Wroclaw
- Russia (2):
  - Cardiology Research Center, Moscow
  - Novosibirsk Research Institute of Circulation Pathology Academician E.N.Meshalkin, Novosibirsk
- Slovak Medical University and National Institute for Cardiovascular Diseases, Bratislava, Slovakia
- Samsung Medical Center, Seoul, South Korea
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitarion 12 Octubre, Madrid
- UniversitätsSpital Zürich, Zurich, Switzerland
- National Taiwan University Hospital, Taipei, Taiwan
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)
- United Kingdom (4):
  - Papworth Hospital, Cambridge
  - Western Infirmary, Glasgow
  - Royal Free London NHS Foundation Trust, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

REFERENCES:
- [Result] Guth S, D'Armini AM, Delcroix M, Nakayama K, Fadel E, Hoole SP, Jenkins DP, Kiely DG, Kim NH, Lang IM, Madani MM, Matsubara H, Ogawa A, Ota-Arakaki JS, Quarck R, Sadushi-Kolici R, Simonneau G, Wiedenroth CB, Yildizeli B, Mayer E, Pepke-Zaba J. Current strategies for managing chronic thromboembolic pulmonary hypertension: results of the worldwide prospective CTEPH Registry. ERJ Open Res. 2021 Aug 16;7(3):00850-2020. doi: 10.1183/23120541.00850-2020. eCollection 2021 Jul. PMID 34409094
- [Derived] Delcroix M, Pepke-Zaba J, D'Armini AM, Fadel E, Guth S, Hoole SP, Jenkins DP, Kiely DG, Kim NH, Madani MM, Matsubara H, Nakayama K, Ogawa A, Ota-Arakaki JS, Quarck R, Sadushi-Kolici R, Simonneau G, Wiedenroth CB, Yildizeli B, Mayer E, Lang IM. Worldwide CTEPH Registry: Long-Term Outcomes With Pulmonary Endarterectomy, Balloon Pulmonary Angioplasty, and Medical Therapy. Circulation. 2024 Oct 22;150(17):1354-1365. doi: 10.1161/CIRCULATIONAHA.124.068610. Epub 2024 Sep 17. PMID 39286890
- See also: Description of the registry on the website of the International CTEPH Association — https://www.cteph-association.org/new-international-cteph-registry.html
- See also: Abstract on long-term outcomes presented at ERS 2021 — https://erj.ersjournals.com/content/58/suppl_65/OA174